CLINICAL TRIAL: NCT01544569
Title: Endogenous DNA Transposition in Rhabdoid Tumors
Brief Title: Studying Biomarkers in Samples From Young Patients With Rhabdoid Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B3; COG-AREN12B3 (Other: Children's Oncology Group); CDR0000727229 (Other: Clinical Trials.gov); AREN12B3 (Other: Children's Oncology Group); NCI-2012-00689 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Cancer
Keywords: rhabdoid tumor of the kidney
MeSH Terms: conditions — Kidney Neoplasms | interventions — In Situ Hybridization, Fluorescence; Gene Expression Profiling; Chromosome Mapping; Microarray Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: gene mapping
Genetic: microarray analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of tissue from patients with rhabdoid tumors in the laboratory may help doctor learn more about changes that occur in DNA and identify genes related to cancer.

PURPOSE: This research trial studies biomarkers in samples from young patients with rhabdoid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the expression and function of transposons in 50 primary rhabdoid tumors.

OUTLINE: Freshly frozen rhabdoid tumors will be studied using fluorescence in situ hybridization (FISH) and polymerase chain reaction (PCR) to establish the genomic location of transposons. Protein expression in rhabdoid tumor tissue microarrays is also analyzed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Freshly frozen rhabdoid tumors from either renal or extra-renal sites from children younger than 2 years of age
* Clinical patient information (age, gender, comorbidities, tumor stage, size, pathology, therapy, outcome) available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: rhabdoid tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Expression and function of transposons in rhabdoid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Mullen, MD, Principal Investigator — Dana-Farber Cancer Institute